CLINICAL TRIAL: NCT06882239
Title: SPINEPASS: SPINE Self-management Techniques for Persistent Headache After Concussion: Physical Therapy Targeting Autonomic and Dura Mater Function
Acronym: SPINEPASS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Queensland (Other)
Collaborators: Brooke Army Medical Center (U.S. Federal Agency); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Dr Lucy Thomas, Principal Investigator, The University of Queensland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HT94252410891; CDMRP-TP230313 (Other Grant/Funding Number: DoD Congressionally Directed Medical Research Program: CDMRP)
Record Dates: First submitted 2025-02-17; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-02

CONDITIONS: Persistent Post-concussive Symptoms; Post Traumatic Headache
Keywords: Persistent post-concussion headache; autonomic; dura; physical therapy; concussion; military
MeSH Terms: conditions — Post-Traumatic Headache; Brain Concussion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SPINEPASS (Experimental): The treatment utilizes anatomy and biomechanics education to inform manual therapy and specific exercises to target areas, such as occipito-atlantal and/or atlanto-axial segmental guarded hypermobility. It also addresses general spinal (thoracic, sacroiliac, rib) and adjacent dysfunction (e.g., temporomandibular joint and lower limb) as required. The treatment targets will be individualized based on initial and ongoing evaluation and will include knowledge, skills, and volitional ingredients. SPINEPASS consists of a core set of three daily exercises integrated into daily activities to improve/restore overall spinal and dural mobility and or stability. It also provides training in the use of specific tools to be used as needed to address symptoms as they occur. Treatment can also include spinal manual therapy and other exercises to enhance the tools, but the emphasis is on self-management.
  Interventions: Other: SPINEPASS Physical Therapy
- Standard Physical Therapy (Active Comparator): Participants will be evaluated by the treating physical therapist to address impairments or dysfunction in cervical musculoskeletal structures, the vestibular and or oculomotor system, and the autonomic nervous system (ANS). They will then be prescribed suitable therapeutic exercises for any cervical, vestibular or oculomotor impairments, and they will be provided with advice and education for graded aerobic exercise and or relaxation and breathing exercises (based on patient preference), consistent with the current recommendations for ANS management post mTBI. The cervical therapy for standard Physical Therapy will be based on impairments found but could include cervical and or thoracic manual therapy, exercises to improve segmental range of motion, exercises for cervical and axioscapular neuromotor retraining, and specific cervical related sensorimotor control exercises such as proprioceptive retraining. A home program of exercises tailored for the individual will be provided.
  Interventions: Other: Standard Physical Therapy

INTERVENTIONS:
Other: SPINEPASS Physical Therapy — SPINEPASS consists of a core set of three daily exercises integrated into daily activities to improve/restore overall spinal and dural mobility and or stability. It also provides training in the use of specific tools to be used as needed to address symptoms as they occur. Treatment can also include spinal manual therapy and other exercises to enhance the tools, but the emphasis is on self-management.
  Arms: SPINEPASS
Other: Standard Physical Therapy — The cervical therapy for standard Physical Therapy will be based on impairments found but could include cervical and or thoracic manual therapy, exercises to improve segmental range of motion, exercises for cervical and axioscapular neuromotor retraining, and specific cervical related sensorimotor control exercises such as proprioceptive retraining. A home program of exercises tailored for the individual will be provided.
  Arms: Standard Physical Therapy

SUMMARY:
This is a prospective randomized controlled trial comparing two different physical therapy approaches to the treatment of posttraumatic headache with autonomic symptoms. AIM 1: To establish the efficacy of SPINEPASS against Standard Physical Therapy to reduce headache disability and impact amongst patients with persistent post-concussion headache. AIM 2: Demonstrate the superiority of SPINEPASS in the efficient self-management of headache. Demonstrate its appropriateness, acceptability, and feasibility and gain patient insights among patients with PPTH compared to standard PT.

DETAILED DESCRIPTION:
Persistent post traumatic headache (PPTH) is a significant problem for the US military affecting up to 33% of service members with a history of mild traumatic brain injury (mTBI) and treatment is usually ineffective. The persistent and chronic nature of PPTH leads to significant disability, burden and reduced readiness. It is commonly migraine-like and associated with visual complaints, and transient neurological abnormalities that can be classified as autonomic nervous system (ANS) in nature. Due to the forces involved during concussion, injury to the brain and neck likely co-occur. Recent research suggests that upper cervical hypermobility may trigger an ANS response and be related to these headaches, due to close anatomical connections to the ANS and dura. Specifically, the dura has unique upper cervical myodural connections to help protect the spinal cord during head movements, with attachments throughout the entire spine. It is innervated by the ANS, is pain sensitive and can cause headache.

The investigators developed a rehabilitation approach to effectively address headache and ANS symptoms in patients. The treatment is hypothesized to influence dura mater and ANS function by addressing the consequences of upper cervical hypermobility. The treatment is a pragmatic biomechanical approach individualized to patients' specific impairments. The approach to this treatment is named SPINE self-management techniques for Persistent headache After concuSSion (SPINEPASS), and it pairs specific personal physical therapy (PT) targets with treatment ingredients.

In this study the investigators plan to conduct a randomized controlled trial (RCT), with a community-based participatory research approach, to explore the efficacy of the SPINEPASS approach on headache disability and self-confidence to manage headache without abortive medication, compared to standard physical therapy (PT) for persistent symptoms post-mTBI. Standard PT will specifically address the neck and the vestibular and oculomotor systems as well as prescribing graded exercise and or relaxation training for management of ANS dysfunction. It does not address the dura mater and while it will aim to stabilize the upper cervical spine, it does not consider the precise restoration of balance of the upper cervical muscles or consider the role of the dura mater to protect and maintain patency of the spinal cord and brain. The investigators will also explore patient experiences and acceptability and feasibility of the program. The hypothesis is that overall, patients will have unique insights and will rate SPINEPASS more appropriate, acceptable and feasible.

Concurrently, the study will include a qualitative arm interviewing participants post-treatment to incorporate an understanding of participants' perspectives on the program to enable effective and sustainable translation of the program into clinical practice. It will consider whether individual confidence for self-management of PPTH is improved in the short and intermediate term and consider participants' perspectives on feasibility, acceptability, and appropriateness of the program as well as factors contributing to the success or failure of these treatment approaches.

Objectives/Specific Aims/Hypotheses:

The purpose of this study is to determine the effect of SPINEPASS, a pragmatic novel PT management program directed towards the spine to target ANS and dura function, in military personnel to reduce headache disability in the short and intermediate term.

The overall objectives of the study are:

1. To test SPINEPASS against standard PT in a randomized controlled trial, (RCT), to improve headache disability.
2. To understand participants' views on the program compared to standard PT and understand factors contributing to success or failure of these treatment approaches. This will be achieved by evaluating patient self-confidence to manage headache, participants' perceptions of the appropriateness, acceptability, and feasibility of SPINEPASS compared to standard PT, and interviewing the participants.

Specific aims and study design:

To evaluate up to 12 sessions of SPINEPASS versus standard PT within a 4- month period and understand participants' views on the program.

Aim 1: Establish the efficacy of the novel, patient centered SPINEPASS against standard PT to reduce headache disability, severity, and impact among patients with PPTH following mTBI using an RCT with a parallel design.

Hypothesis 1.1a: Individuals with PPTH will have significant improvement in headache disability (HIT-6) (primary outcome) following SPINEPASS compared to those who have standard PT immediately following treatment [Primary outcome].

Hypothesis 1.1b: Participants who undergo SPINEPASS will have significantly greater improvements in headache severity (i.e., intensity range, frequency, duration, medication intake), related symptom severity (i.e., autonomic symptom severity), and functional outcomes (i.e., self-efficacy, quality of life, health locus of control) compared to standard PT [secondary outcomes].

Hypothesis 1.2: Participants who complete SPINEPASS will continue to report significantly less headache disability than those who complete standard PT at the 3 and 12-month follow-up [T2 and T3].

Aim 2: Demonstrate the superiority of SPINEPASS in the efficient self-management of headache and, in its appropriateness, acceptability, and feasibility and patient insights among patients with PPTH compared to standard PT.

Hypothesis 2.1: Individuals with PPTH will have significant improvement in self-confidence to manage headache (a) lower intensity and b) eliminate entirely) without abortive medication at T1, T2, T3 following SPINEPASS compared to those who have standard PT.

Hypothesis 2.2: Patients who undergo SPINEPASS will require fewer treatment sessions to achieve 50% confidence to manage (lower and or eliminate) headaches without abortive medication and fewer treatments overall compared to the standard PT group.

Hypothesis 2.3: Participants in SPINEPASS will have better adherence to the exercise program compared to Standard PT.

Hypothesis 2.4: Participants will find the SPINEPASS program appropriate, acceptable, and feasible on quantitative measures (Appropriateness of Intervention, Acceptability of Intervention, Feasibility of Intervention measures).

Hypothesis 2.5: Participants will have unique insights into factors contributing to the success or failure of the individual treatment approaches and home exercises compatible with military lifestyle [themes from qualitative interview].

ELIGIBILITY:
Inclusion Criteria:

* Persistent Post-traumatic headache (PPTH) duration =or > 4 weeks.
* No self-reported improvement in headache pattern in the past 3 weeks. (Patients will be asked to determine whether the usual pattern of their headaches has changed for the better over the last 3 weeks.
* Compass-31 score > 21 to select patients who have evidence of ANS dysfunction which SPINEPASS aims to address.
* Headache Impact Test (HIT6) =>50 to capture headache-related disability of "some impact" or more.
* Headache worst intensity >3/10 on a numerical rating scale (NRS), at least once per week.

Exclusion Criteria:

* Contraindications for spinal or graded general exercise.

  * Contraindications to spinal manual therapy at or below C5-6 level
* Cognitive impairment/ language barriers affecting ability to participate.
* Redeployment/relocation or retirement planned within the next 6 months to reduce the chances of dropouts to treatment and follow-up.
* Rating self-confidence to manage (eliminate and or lower) headaches without abortive medication at baseline of 30% or greater.
* Inability to attend up to 12 in-person treatment sessions for 4 months.
* Unwilling to limit commencement of other management for PPTH during the trial period.
* Botox for headache management within the last 8 weeks or during the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2028-03-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Headache Impact Test (HIT-6) | Baseline to T1 (treatment completion -up to 12 weeks), T2 (3 months following T1), T3 (12 months following T1)
  The HIT-6 is a validated measure of disability associated with headache and has been shown to be useful in migraine. A higher score indicates greater disability. Scores between 50 and 55 represent some impact; scores between 56 and 59 represent substantial impact, and scores > 60 indicate severe impact. A reduction in the score of six or more is considered a clinically meaningful change.
Confidence to self-manage headache | Baseline; T1 (treatment completion- up to 12 weeks); T2 (3 months post T1)
  An electronic diary will ask the patients to rate their perceived ability to self-manage (a) lower and b) eliminate their headache using the exercises or tools, (without abortive medication measures), each week using a % scale, where 100% indicates the patient can manage it perfectly and 0% indicates an inability to manage the headache. This score is based on measures of global perceived effect or rating scales but modified to be captured in a percentage score.

SECONDARY OUTCOMES:
Composite Autonomic Symptom Score (COMPASS-31) | Baseline to T1 (treatment completion -up to 12 weeks), T2 (3 months following T1), T3 (12 months following T1)
  COMPASS-31) is a validated measure and quantifies 6 domains relating to ANS function: orthostatic intolerance, vasomotor, secretomotor, gastrointestinal, bladder and pupillomotor. The 6 subscales are weighted and sum to a total COMPASS-31 score of 0 to 100 with higher scores indicating greater disability. Medians and ranges for healthy volunteers are 10 ± 8 (mean age 46.6 years). Scores of >21 indicate elevated autonomic symptoms. Usually the score is based on symptoms in the year preceding assessment. To allow comparison of symptoms during treatment we have investigated using a modified version of the questionnaire for symptoms over the last month and compared it to the original questionnaire (last year). The COMPASS-31 (last month) was comparable (last year), and the COMPASS-31 (last month) was responsive with a large effect size (1.3) post-intervention, suggesting that this is a suitable outcome measure for use in these participants.
Neurobehavioral Symptom Inventory (NSI). | Baseline to T1 (treatment completion -up to 12 weeks), T2 (3 months following T1), T3 (12 months following T1)
  The NSI is a 22-item inventory/88 that assesses symptoms associated with TBI with established reliability and validity, although these symptoms are not specific to concussion. Responses range from 0 (none) to 4 (very severe) and address how much each symptom has disturbed the patient in the last two weeks.43, 44 This documents patients' subjective complaints across ocular, vestibular/auditory, cognitive, and affective domains. Both total and domain scores will be used to document the characteristics of the cohort as this measure is routinely used in the US military following TBI.

CONTACTS AND LOCATIONS:
Overall Officials: Lucy C Dr Lucy Thomas, PhD, Principal Investigator — The University of Queensland; Julia M Dr Julia Treleaven, PhD, Principal Investigator — University of Queensalnd; Amy 0 Dr Amy Bowles, MD, Study Director — Brooke Army Medical Center
Locations (1):
- Brook Army Medical Center, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD will be provided to FITBIR. The Department of Defense, in collaboration with the National Institutes of Health, has developed the Federal Interagency Traumatic Brain Injury Research (FITBIR) Informatics System, a central repository and resource for sharing data to promote collaboration, accelerate research, and advance knowledge on the characterization, prevention, diagnosis, and treatment of TBI. FITBIR provides a common platform and standardized format for data collection, retrieval and archiving, while allowing for flexibility in data entry and analysis.
Time Frame: IPD will be provided to FITBIR on an annual basis for 4 years starting in 01 October 2025 to 01 October 2028.
Access Criteria: Other researchers conducting research in traumatic brain injury and registered with FITBIR will be able to access de-identified IPD from the study.
URL: https://fitbir.nih.gov/

REFERENCES:
- [Background] Patricios JS, Schneider KJ, Dvorak J, Ahmed OH, Blauwet C, Cantu RC, Davis GA, Echemendia RJ, Makdissi M, McNamee M, Broglio S, Emery CA, Feddermann-Demont N, Fuller GW, Giza CC, Guskiewicz KM, Hainline B, Iverson GL, Kutcher JS, Leddy JJ, Maddocks D, Manley G, McCrea M, Purcell LK, Putukian M, Sato H, Tuominen MP, Turner M, Yeates KO, Herring SA, Meeuwisse W. Consensus statement on concussion in sport: the 6th International Conference on Concussion in Sport-Amsterdam, October 2022. Br J Sports Med. 2023 Jun;57(11):695-711. doi: 10.1136/bjsports-2023-106898. PMID 37316210
- [Background] Schneider KJ, Critchley ML, Anderson V, Davis GA, Debert CT, Feddermann-Demont N, Gagnon I, Guskiewicz KM, Hayden KA, Herring S, Johnstone C, Makdissi M, Master CL, Moser RS, Patricios JS, Register-Mihalik JK, Ronksley PE, Silverberg ND, Yeates KO. Targeted interventions and their effect on recovery in children, adolescents and adults who have sustained a sport-related concussion: a systematic review. Br J Sports Med. 2023 Jun;57(12):771-779. doi: 10.1136/bjsports-2022-106685. PMID 37316188
- [Background] Bartsch T, Goadsby PJ. Increased responses in trigeminocervical nociceptive neurons to cervical input after stimulation of the dura mater. Brain. 2003 Aug;126(Pt 8):1801-13. doi: 10.1093/brain/awg190. Epub 2003 Jun 23. PMID 12821523
- [Background] Sillevis R, Hogg R. Anatomy and clinical relevance of sub occipital soft tissue connections with the dura mater in the upper cervical spine. PeerJ. 2020 Aug 10;8:e9716. doi: 10.7717/peerj.9716. eCollection 2020. PMID 32864219
- [Background] Fazliogullari Z, Kilic C, Karabulut AK, Yazar F. A morphometric analysis of the superior cervical ganglion and its surrounding structures. Surg Radiol Anat. 2016 Apr;38(3):299-302. doi: 10.1007/s00276-015-1551-3. Epub 2015 Sep 12. PMID 26364034
- [Background] Esterov D, Greenwald BD. Autonomic Dysfunction after Mild Traumatic Brain Injury. Brain Sci. 2017 Aug 11;7(8):100. doi: 10.3390/brainsci7080100. PMID 28800081
- [Background] Howard L, Dumkrieger G, Chong CD, Ross K, Berisha V, Schwedt TJ. Symptoms of Autonomic Dysfunction Among Those With Persistent Posttraumatic Headache Attributed to Mild Traumatic Brain Injury: A Comparison to Migraine and Healthy Controls. Headache. 2018 Oct;58(9):1397-1407. doi: 10.1111/head.13396. Epub 2018 Aug 29. PMID 30156267
- [Background] Goodrich GL, Flyg HM, Kirby JE, Chang CY, Martinsen GL. Mechanisms of TBI and visual consequences in military and veteran populations. Optom Vis Sci. 2013 Feb;90(2):105-12. doi: 10.1097/OPX.0b013e31827f15a1. PMID 23314131